CLINICAL TRIAL: NCT04727697
Title: Patient Reported Outcomes, Satisfaction, and Understanding Following Orthopaedic Ambulatory Procedures Using Augmented/Virtual Reality as an Education Tool
Brief Title: Augmented Reality Perioperative Training and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Lee Kaplan, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20201439
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care, preoperative teaching group (Active Comparator): The participants in this group will receive the preoperative teaching and handouts as is the current standard of care.
  Interventions: Other: Standard of Care preoperative teaching and handouts
- Augmented Reality perioperative experiences group (Experimental): The participants in this group will receive the preoperative teaching and handouts as is the current standard of care in addition to receiving the augmented reality (AR) perioperative experience.
  Interventions: Other: Augmented Reality; Other: Standard of Care preoperative teaching and handouts

INTERVENTIONS:
Other: Augmented Reality — Patients will receive the preoperative AR experience during their immediately preoperative office visit. The duration of the exposure is approximately 15 minutes.
  Arms: Augmented Reality perioperative experiences group
Other: Standard of Care preoperative teaching and handouts — At preoperative appointments, patients receive verbal teaching and written handouts about day of surgery instructions and expectations.

SUMMARY:
The purpose of this study is to learn more about how augmented reality systems can influence perioperative experience and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years old or greater
* Patients who have a scheduled ambulatory procedure with University of Miami Orthopaedic providers.

Exclusion Criteria:

* Any patient not scheduled for procedures
* Minors
* Cognitively incapacitated
* Prisoners.
* Have any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the patient from meeting or performing study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety as measured by the state-trait anxiety inventory (STAI) | Baseline, up to 14 days
  STAI has scores ranging from 20 to 80 with higher scores corresponding to greater levels of anxiety.

SECONDARY OUTCOMES:
Change in comfort level as measured by perioperative comfort questionnaire | Baseline, up to 14 days
  Perioperative comfort questionnaire ranges from 1-5 with higher scores indicating greater levels of comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Kaplan, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rizzo MG Jr, Costello JP 2nd, Luxenburg D, Cohen JL, Alberti N, Kaplan LD. Augmented Reality for Perioperative Anxiety in Patients Undergoing Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2023 Aug 1;6(8):e2329310. doi: 10.1001/jamanetworkopen.2023.29310. PMID 37589975